CLINICAL TRIAL: NCT03214315
Title: Réseau Structurant Sur le Cancer de la Prostate du Grand Ouest
Brief Title: Structural Network on Prostate Cancer in the French Greater West Region
Acronym: RESCAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Nantes University Hospital (Other); Rennes University Hospital (Other); University Hospital, Angers (Other Government); Poitiers University Hospital (Other); Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: AOCGO13-GF-RESCAP; DC-2014-2045 (Registry Identifier: CPP)
Record Dates: First submitted 2017-06-26; First posted 2017-07-11 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample of visceral adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostatectomy: Visceral adipose tissue specimen sample
  Interventions: Procedure: Visceral adipose tissue specimen

INTERVENTIONS:
Procedure: Visceral adipose tissue specimen — specimen
  Other Names: specimen

SUMMARY:
The project aims at developing and structuring a network of clinicians, pathologists, and scientists, from the "Grand Ouest" area, most of them already involved in prostate cancer management and research.

Patients treated by radical prostatectomy will be recruited within the ReSCaP network of clinicians, with centralized database and standardized bio-resource collection, including prostate and adipose tissue samples. Seven clinical centers will participate to the network, 6 recruiting mainly Caucasian patients, and 1 from the French West Indies recruiting mainly African Caribbean patients. After 18 months, 1000 patients will be included.

The main goal is to study the relationships between adipose tissue/lipids and prostate cancer aggressiveness. In fact, adipose tissue is likely to be involved in cancer progression at many levels: abdominal obesity has been associated with aggressive disease, and poly-unsaturated fatty acids (PUFAs), as well as cytokines produced by adipocytes (adipokines) have an impact on cancer cells growth and migration in vitro. Moreover, adipose tissue is the preferential site of storage of persistent organic pollutants with estrogenic properties, which could impact cancer progression.

The study will analyze the association between adipose tissue (distant from the prostate) composition and cancer aggressiveness. Among the 1000 patients, 100 aggressive tumors will be selected according to the d'Amico criteria (Gleason score 8 or more and/or pT3 tumors). They will be matched with 100 potentially indolent prostate cancers (Gleason 6 or less, and PSA less than 10, and pT2 stage on the surgical specimen). These 200 adipose tissue samples will be analyzed for 1/ the lipid profile, including the fatty acid composition, particularly PUFAs, that reflects past dietary fat intake, 2/ adipokine expression, and 3/ tissue concentrations of persistent organic pollutants belonging to the class of organochlorine pesticides with hormone-like activity.

DETAILED DESCRIPTION:
Relevance and strategic approach Prostate Cancer (PCa) is the most common cancer in men and the second leading cause of cancer deaths in western countries. Known risk factors are advanced age, ethnic origins and positive family history of the disease (1). There are considerable ethnic disparities in PCa risk, with a 60% higher incidence rate among African-American (AA) men as compared with European-American (EA) men (2). Similarly, in the French West Indies, where at least 90% of inhabitants are of African descent, the incidence of PCa is twice as high as in the rest of France (3). Many lifestyles, environmental and occupational related risk factors including obesity, diet, medications and pesticides have been implicated in PCa etiology, but their roles remain unclear (4). Current research suggests that there is a complex interplay of genetic and environmental factors that have a causative role in PCa.

PCa also has a highly heterogeneous potential of evolution. While some cancers will behave in an aggressive manner, other patients will have an indolent form of the disease that could not require any treatment. Several parameters are used to predict the risk of evolution in PCa patients, either before any treatment: clinical stage, Gleason score on biopsies, and serum prostatic specific antigen (PSA), or after the analysis of radical prostatectomy specimens: pathological stage and surgical Gleason score (5). However, despite the value of these prognostic factors, the potential of aggressiveness remains difficult to assess at diagnosis, and patients classified within the intermediate risk group are often difficult to manageThere is a challenge to discover new markers and novel targets for early therapeutic manipulation.

Both genetic and environmental factors have been linked to the risk of aggressive disease. The ethnic origin is likely to play a role, since the proportion of cases diagnosed at the metastatic stage is reported to be higher for African-American patients (35%) than for European-American patients (22%), with a 2.4-fold higher mortality rate in AA men than in EA men (2).Together with genetic factors, environmental factors also seem to play a key role in PCa progression. Some environmental factors such as obesity have been associated with aggressive PCa (6). However, much remains to search about the role of genetic and environmental factors and their interplay in PCa aggressiveness. White adipose tissue (WAT) and lipids are potentially involved in the development and/or progression of PCa at many levels.

WAT is a metabolically active endocrine organ. Adipocytes secrete a variety of hormones, bioactive peptides and cytokines, termed adipokines (9). Several adipokines have been involved in the mechanisms leading to PCa progression and aggressiveness, including leptin, interleukin IL-6 and vascular endothelial growth factor (VEGF).

Storage of endocrine disruptors. Endocrine disruptors (ED) are thought to be involved in prostate cancer (10). However, epidemiologic evidence of a positive link between environmental exposures to ED is limited. Two studies using blood plasma or abdominal fat for monitoring persistent pollutants have shown positive associations with PCa risk (transchlordane, beta-hexachlorocyclohexane, trans-nonachlore, dieldrine, and polychlorinated biphenyl 153) (11, 12). A recent study carried out in French West Indies showed that chlordecone, an organochlorine pesticide with well defined estrogenic properties, increases the risk of PCa, and is associated with an aggressive form of the disease in subjects with a positive family history of PCa (13).

WAT composition: Lipidome. Among nutrients, dietary lipids are major determinants of the overall lipid composition of WAT, as assessed during dietary intervention studies (19-22). Among fatty acids, essential polyunsaturated fatty acids (PUFAs) are a subclass of bioactive components divided in two groups, n-6 and n-3 fatty acids. The n-6 series include the precursor linoleic acid (LA, 18:2n-6). The n-3 series include the precursor alpha-linolenic acid (ALA, 18:3n-3), and highly unsaturated derivatives. The fatty acid composition of WAT has been shown to reflect the past fatty acid intake (23). Although there are no conclusive studies showing an association between total dietary fat intake and PCa risk, specific types of dietary fat (animal fat) appear to be more significant in increasing PCa risk (6, 28). The association between fish consumption (rich in in the long-chain omega-3 PUFAs) and lower risk of prostate cancer is controversial, but a significant reduction in prostate cancer-specific mortality has been described (29). Previous studies analyzing the PUFAs composition in prostate tissues have led to conflicting results. However, fatty acid composition of WAT has never been studied in PCa in association with aggressiveness and progression.

The objective of the program is to structure a network associating clinicians, pathologists, and scientists devoted to prostate cancer management and research. The network will generate a multi-centric centralized database of PCa patients treated by radical prostatectomy, with standardized bio-resources collection, including prostate and adipose tissue samples. The use of the bio-resources will be orientated mainly toward the relationships between adipose tissue/lipids and PCa aggressiveness.

The project aims to characterize an association between PCa aggressiveness and the composition of pelvic adipose tissue. Adipose tissue samples from patients with either low risk (n=100) or aggressive (n=100) PCa will be analyzed for 1/ the lipid profile (fatty acid composition and phospholipids proportions), 2/ expression of adipokines, and 3/ persistent organic pollutants with hormone-like activity. The analysis will take into account known factors of aggressiveness, including obesity, MetS components, ethno-geographic origin, and positive family history of the disease.

Methodology and techniques implemented I- Constitution of the database and bio-resources collection Each patient with prostate cancer treated by radical prostatectomy in the 7 clinical centers of the network will be included in the cohort. Given the surgical activity of these centers during the last 3 years, a minimum of 1000 inclusions is expected after 18 months, with around 250 african-carribean patients.Standardized clinical, biological, and pathological data will be entered in a common centralized eCRF available in each center (Clinsight®) with central management and validation (Team 13). Financial support will be provided to the clinical teams for entering the data (technicians specialized in clinical research).

The data commonly associated with PCa will be entered in the database: administrative items (name, DOB, address, Hospital N°, Pathology N°), preoperative PSA, clinical stage, pathological items (weight and size of the specimen, pathological stage including lymph node status, Gleason score, % of grade 4 ou 5, greater axis of the main focus, margin status), and follow-up items (both biological and clinical).The following items will also be specified: BMI, waist circumference, fasting glucose, blood pressure, circulating lipids (triglycerides, total, LDL and HDL cholesterol), ongoing treatments (lipid lowering drugs, HTA, treatments for diabetes), ethno-geographic origin, and family history of PCa During the surgical procedures, 3 pieces of pelvic adipose tissue (around 5g, 2g and 2 g, for tasks 1, 2, and 3 of Axis 1, respectively) will be sampled, sent to the biological resource center, and immediately frozen at -80°C. The investigators choose to sample visceral WAT instead of subcutaneous WAT, because visceral adipocytes are more metabolically active (8). Among visceral WAT, the investigators choose to sample perivesical adipose tissue, since fat around the bladder is always very abundant, and can be easily taken during the surgical procedure. The prostate specimens will be sent immediately to the pathology departments, and managed in a standardized manner.

The patients included in the cohort will be asked to sign an informed consent (after agreement of the Ethical Committee/IRB). The annotated bio-resources concerning the subjects included in the programs will be managed in respect of the rules defined by the CNIL.

Selection of patients with either aggressive or low risk disease from the cohort from the 1000 patients expected at M18, 100 patients with highly aggressive disease will be selected. Selection will be made based on the criteria of high risk disease, mainly high grade PCa (Gleason score 8 or more) and/or pathological stage pT3. Each of these 100 patients will then be matched (center by center) with 1 patient with indolent disease and identical status for age (50 or less, 51-55, 56-60, 61-65, 66-70, 71-75, more than 75 years old) and BMI (normal, overweight, and obese). Criteria for indolent disease will include preoperative PSA < 10ng/ml, and Gleason score 6 or less (on the surgical specimen), and pT2 stage. If several indolent cases could be matched with 1 aggressive case, the one with the smaller tumor size will be preferred. Adipose tissue sampled from these 200 patients will be used.

The aim is to identify associations between aggressive and significant PCa and the composition of adipose tissue. The investigators hypothesize that persistent organic pollutants (that reflect cumulative past exposure), and/or lipid composition (that reflect past intake), could be, together with adipokines expression, associated with disease aggressiveness. Known factors of PCa aggressiveness (ethnic origin, familial history, and obesity status) will be taken into account.

Task1: Lipidome analysis Analyses performed on the adipose tissue samples will be: i) triglyceride fatty acid composition, and ii) adipose cells membrane phospholipids classes relative amounts. Five major phospholipids classes found in the plasma membrane of adipose cells can be separated and quantified: phosphatidylcholine, phosphatidylethanolamine, phosphatidylinositol, phosphatidylserine and sphingomyelin. Adipose tissue being mostly composed of triacylglycerol and only approximately 1% phospholipids, the study of membrane phospholipids will require larger sample amounts (5 g) than would typically be necessary for triglycerides fatty acid composition analysis (400-500 mg).

Adipose tissue samples will undergo lipid extraction with the use of chloroform and methanol (according to the Folch method). Briefly, total extract will be vacuum-dried, then resolubilized in a mixture of hexane and methanol to partition neutral (hexane soluble) and polar (methanol soluble) lipids. Triglycerides in the hexane phase will be further purified from other neutral or polar lipids by thin layer chromatography on silica-gel plates. Purified triglycerides will undergo methanol transesterification to produce volatile fatty acids as methyl esters. Separation and quantification of fatty acids will be performed by gas chromatography (BPX-70 phase capillary column, on-column injection, flame-ionization detector).

Task2: Adipokine measurements Total RNA from adipose tissue samples will be extracted by the Trizol technique and RNA quality will be checked by gel agarose electrophoresis and quantification by NanoDrop. After reverse transcription of encoding mRNA into cDNA, control quality of reverse transcription PCR amplification will be done using a housekeeping gene in the low number of cycles and new control by gel agarose. Real-time quantitative PCR will then be performed in triplicate on nine genes of interest (adipokines) and three housekeeping genes for normalization (18S, beta-actin and SDHA), ie 10 800 points generated. PCRs will be made in 384-well plates and the reaction mixtures distributed by robot distribution.Adipokine list (n=9): chemerin, interleukin-6 (IL-6), plasminogen activator inhibitor-1 (PAI-1), retinol binding protein 4 (RBP4), tumor necrosis factor-alpha (TNF alpha), visfatin, leptin, adiponectin, apelin.

Task3: Measurements of persistent organic pollutants (organochlorine pesticides) The analytical methodology used for measuring the targeted organochorine pesticides is derived from procedures previously developed, validated, and accredited for other classes of lipophilic persistent organic pollutants such as dioxins and PCB compounds. Briefly, a preliminary step using accelerated solvent extraction (ASE) will be followed by successive purification stages on activated silica and celite columns. The measurement will be performed using gas chromatography coupled to high resolution and/or tandem mass spectrometry (GC-HRMS, GC-MS/MS). The quantification will be achieved according to the isotopic dilution method (i.e. using 13C labeled analogous as internal standards). The selection of the main targeted substances will be preliminary based on the Stockholm convention that lists about 12 major pesticides of concern.

The multicenter standardized clinical and biological database will identify 2 homogeneous groups of PCa patients with characteristics of either aggressive or potentially indolent disease. The investigators expect that the analysis of pelvic adipose tissue will demonstrate whether some categories of 1/ Lipids (reflecting the diet), 2/ Adipokines and 3/ Stored Xenobiotics are preferentially associated with a greater or lower risk of PCa aggressiveness. Such identification could then lead to preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for prostate cancer by radical prostatectomy without previous therapy
* Informed written consent

Exclusion Criteria:

• Subject to deprivation of liberty, under guardianship or guardianship, under safeguard of justice, minor or major inability to express his or her consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients treated for prostate cancer by radical prostatectomy
Study Population: Patients treated for prostate cancer by radical prostatectomy in the 7 university hospital partners of the study
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
Dietary intake of essential fatty acids | Participant exposure from birth until diagnosis date of Prostate Cancer
  Past dietary intake of essential fatty acids is quantified by measuring their concentration in white adipose tissue

SECONDARY OUTCOMES:
Exposure to persistant organic pesticides | Participant exposure from birth until diagnosis date of Prostate Cancer
  Exposure to persistant organic pollutants (organochlorine chemicals, which are fat-soluble) is quantified by measuring the concentration in white adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle FROMONT-HANKARD, MD-PHD, Study Director — University François Rabelais of TOURS
Locations (7):
- France (6):
  - Urology CHRU-TOURS, Tours, I&L
  - University Hospital, Angers
  - University Hospital, Brest
  - University Hospital, Nantes
  - Uniersity Hospital, Poitiers
  - University Hospital, Rennes
- University Hospital, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No